CLINICAL TRIAL: NCT06815965
Title: An Open-Label Phase 2a Clinical Study of the P38 Alpha Kinase Inhibitor Neflamapimod in Patients With Dementia With Lewy Bodies (DLB)
Brief Title: A Clinical Study of Neflamapimod in Patients With Dementia With Lewy Bodies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: CervoMed, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EIP22-NFD-505; 2024-511446-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-23; First posted 2025-02-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Dementia With Lewy Bodies (DLB)
Keywords: Dementia; France; neflamapimod
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — VX-745

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neflamapimod, Open-label (Experimental): Neflamapimod will be administered orally, with food, for 24 weeks in subjects with DLB. Subjects will receive 4 capsules per day (80 mg BID), two capsules in the morning and two capsules in the evening, with food (i.e., with the morning and evening meals)
  Interventions: Drug: neflamapimod

INTERVENTIONS:
Drug: neflamapimod — Neflamapimod is a highly specific inhibitor of the intra-cellular enzyme mitogen-activated protein kinase 14 (p38α). It is administered orally in 40 mg capsules.
  Other Names: VX-745

SUMMARY:
The purpose of this clinical study is to evaluate the safety and tolerability (side effects) and pharmacokinetics (drug levels in the body) of 80mg neflamapimod given twice daily in patients with dementia with Lewy bodies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥55 years.
2. Subject is willing and able to provide written informed consent.
3. Probable DLB by consensus criteria (McKeith et al, 2017; McKeith et al, 2020).
4. MoCA score ≥18 OR CDR global score (CDR-GS) ≤ 1.0 during Screening.
5. If the patient is currently receiving cholinesterase inhibitor and/or memantine therapy, the patient must have received such therapy for greater than 3 months and on a stable dose for at least 6 weeks at the time of enrollment. Except for reducing the dose for tolerability reasons, the dose of cholinesterase inhibitor may not be modified during the study. If the patient is not currently receiving such therapy, but received such therapy previously, that therapy must have been discontinued at least 3 months prior to enrollment.
6. Normal or corrected eyesight and auditory abilities, sufficient to perform all aspects of the cognitive and functional assessments.
7. No history of learning difficulties that may interfere with their ability to complete the cognitive tests.
8. Received vaccination for SARS-CoV-19 unless medical contraindications prevent being vaccinated or has a history of natural infection.
9. Must have reliable informant or caregiver.

Exclusion Criteria:

1. Diagnosis of any other ongoing central nervous system (CNS) condition other than DLB, including, but not limited to, post-stroke dementia, vascular dementia, Alzheimer's disease (AD), Frontotemporal dementia (FTD), or Parkinson's disease (PD).
2. Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
3. Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
4. Diagnosis of alcohol or drug abuse within the previous 2 years.
5. Poorly controlled clinically significant medical illness, such as hypertension (blood pressure >180 mmHg systolic or 100 mmHg diastolic); myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would interfere with assessment of drug safety.
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN), total bilirubin >1.5 × ULN, and/or International Normalized Ratio (INR) >1.5. If patient is taking blood thinners (e.g., warfarin), and has no known liver issues, INR >3.
7. Positive screen for human immunodeficiency virus, hepatitis B surface antigen (HbsAg), antibody (anti-HbS), hepatitis C virus (HCV) antibody or evidence of latent or active tuberculosis, active opportunistic or life-threatening infections.
8. Participated in a study of an investigational drug less than 6 weeks or 5 half-lives of an investigational drug, whichever is longer, before enrollment in this study.
9. Receipt of a live vaccine, with the exception of influenza, within 4 weeks before starting study drug treatment.
10. History of previous neurosurgery to the brain within the past five years.
11. If male with female partner(s) of child-bearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
12. If female who has not has not reached menopause >1 year previously or has not had a hysterectomy or bilateral oophorectomy/salpingo-oophorectomy, has a positive pregnancy test result during Screening and/or is unwilling or unable to adhere to the contraception requirements specified in the protocol.
13. If female, currently pregnant or breastfeeding.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability 80 mg neflamapimod given twice daily in patients with dementia with Lewy bodies. | From enrollment until the end of treatment at 24 weeks
  The safety and tolerability of 80 mg neflamapimod given twice daily in patients with dementia with lewy bodies will be evaluated via the incidence of treatment-emergent Adverse events (AEs) and Serious adverse events (SAEs) during 24 weeks of treatment
Evaluate the safety and tolerability of 80mg neflamapimod given twice daily in patients with dementia with Lewy bodies. | From enrollment until the end of treatment at 24 weeks
  The safety and tolerability of 80 mg neflamapimod given twice daily in patients with dementia with lewy bodies will be evaluated via the incidence of elevations in amino-alanine transferase (ALT) and/or aspartate amino-transferase (AST) ≥ three times the upper limit of normal during 24 weeks of treatment
Evaluate the maximum plasma concentration (Cmax) of 80mg neflamapimod given twice daily in patients with dementia with Lewy bodies. | From enrollment until the end of treatment at 24 weeks
  The maximum plasma concentration (Cmax) of 80 mg neflamapimod given twice daily in patients with dementia with lewy bodies will be evaluated via mean (with 95% confidence interval) plasma drug concentration at steady state during 24 weeks of treatment with neflamapimod 80mg BID.
Evaluate the trough plasma concentration (Ctrough) of 80mg neflamapimod given twice daily in patients with dementia with Lewy bodies. | From enrollment until the end of treatment at 24 weeks
  The trough plasma concentration (Ctrough) of 80 mg neflamapimod given twice daily in patients with dementia with lewy bodies will be evaluated via mean (with 95% confidence interval) plasma drug concentration at steady state during 24 weeks of treatment with neflamapimod 80mg BID.

SECONDARY OUTCOMES:
Change in ADNI-EF composite score from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in the mean composite score for Alzheimer's Disease Neuroimaging Initiative Executive Functioning composite scale (ADNI-EF) from baseline to 24 weeks where composite scores range from -3.0 to 3.0 and a positive change in composite score indicates improvement in cognition and a negative change in composite score indicates a worsening in cognition.
Change in CDR-SB score from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in the Clinical Dementia Rating Sum of Boxes (CDR-SB) score from baseline to 24 weeks. CDR-SB scores range from 0 to 18 with a higher score indicating worsening of cognitive impairment.
Change in TUG test results from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in Timed Up and Go (TUG) test results from baseline to 24 weeks. TUG scores typically range from 6 to 20 seconds with a lower score indicating better mobility and a higher score indicating worse mobility.

OTHER OUTCOMES:
Change in MBI-C score from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in the Mild Behavioral Impairment Checklist (MBI-C) scale from baseline to 24 weeks. The scale ranges from 0 to 102, with lower scores indicating less severe symptoms and higher scores indicating more severe symptoms.
Changes in DCFS from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in the Dementia Cognitive Fluctuations Scale (DCFS) score from baseline to 24 weeks. DCFS scores range from 4 to 20 where a higher score indicates more severe cognitive fluctuations and disease worsening.
Changes hallucinations (PDAP questionnaire) from baseline to 24 weeks | From enrollment until the end of treatment at 24 weeks
  Effects of neflamapimod treatment will be assessed via changes in hallucinations as measured by the Parkinson's disease-associated psychotic symptoms questionnaire (PDAP) score from baseline to 24 weeks where a higher score indicates more severe symptoms. The scores range from 0 to 9 for patient responses and 0 to 9 for caregiver responses where a lower score indicates improvement and a higher score indicates worsening in condition.
Changes in NBM volume from baseline to 16 weeks | From enrollment until 16 weeks
  Effects of neflamapimod treatment will be assessed via changes in volume of nucleus basalis of Meynert (NBM) as measured by structural Magnetic Resonance Imaging (MRI) from baseline to 16 weeks where a reduction in volume indicates degeneration.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Lariboisière - APHP; Centre de Neurologie Cognitive, Paris
  - Strasbourg University Hospital (Les Hopitaux Universitaires de Strasbourg), Strasbourg

IPD SHARING:
Plan to Share IPD: No